CLINICAL TRIAL: NCT02338388
Title: Longitudinal Transvaginal Ultrasound Evaluation of Cesarean-scar Thickness in the First Two Years After Single- or Double-layer Uterotomy Closure: a Prospective Randomized Study
Brief Title: Cesarean-scar Thickness and Closure Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Bamberg (Other)
Responsible Party: Sponsor-Investigator, Christian Bamberg, Christian Bamberg, MD, PhD, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: (EA1/149/11)
Record Dates: First submitted 2015-01-12; First posted 2015-01-14 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Uterine Scar Remodeling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Single-layer unlocked closure (Active Comparator)
  Interventions: Procedure: cesarean section technique
- Single-layer locked closure (Active Comparator)
  Interventions: Procedure: cesarean section technique
- Double-layer closure (Active Comparator): The first layer was continuous and unlocked and a second, continuous non-locking imbricating layer was applied over the first suture.
  Interventions: Procedure: cesarean section technique

INTERVENTIONS:
Procedure: cesarean section technique — Comparing three different types of suturing the uterus at Cesarea section

SUMMARY:
The aim of this trial is the surgical method in cesarean deliveries, especially the uterotomy closure technique.

DETAILED DESCRIPTION:
The aim of this prospective, randomized controlled trial was to longitudinally evaluate uterine-scar remodeling via transvaginal ultrasound after single- or double-layer uterine closure six weeks and at least six months after Cesarean delivery.

The women were included at their booking visit for an elective CD or during labor before an nonemergent CD. They were randomly assigned for three different uterotomy suture techniques: The uterus was closed with a continuous single layer locked stitch or continuous single unlocked layer or double layer.

Six weeks and between six and twenty-four month after their cesarean delivery the women were examined by transvaginal ultrasound with an empty maternal bladder, in a supine decubitus position using a GE E8 system equipped with a 5-9 MHz transducer (GE Healthcare, Milwaukee, WI).

The measurement of the uterine scar thickness was performed perpendicular to the uterine wall and was defined as shortest visible distance between the decidua and the delineation of the endometrium at the level of the cesarean scar.

ELIGIBILITY:
Inclusion Criteria:

* Elective cesarean section
* Cesarean section during labor

Exclusion Criteria:

* Emergency cesarean section
* Declined to participate

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2012-01; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
cesarean scar-thickness | 24 months

REFERENCES:
- [Derived] Bamberg C, Hinkson L, Dudenhausen JW, Bujak V, Kalache KD, Henrich W. Longitudinal transvaginal ultrasound evaluation of cesarean scar niche incidence and depth in the first two years after single- or double-layer uterotomy closure: a randomized controlled trial. Acta Obstet Gynecol Scand. 2017 Dec;96(12):1484-1489. doi: 10.1111/aogs.13213. Epub 2017 Sep 21. PMID 28832909